CLINICAL TRIAL: NCT00712140
Title: Persephone: Duration of Trastuzumab With Chemotherapy in Women With Early Stage Breast Cancer: Six Months Versus Twelve
Brief Title: Trastuzumab in Treating Women With HER2-Positive Early Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Warwick Medical School (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000598391; WMS-PERSEPHONE; MREC-PERSEPHONE; EUDRACT: 2006-007018-39; ISRCTN 52968807; MREC 07/MRE08/35; EU-20858; CRUK-BRD/07/137
Record Dates: First submitted 2008-07-08; First posted 2008-07-09 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2008-11

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

ARMS (2):
- Arm I (Active Comparator): Patients receive trastuzumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 12 months in the absence of disease progression or unacceptable toxicity. All patients also receive standard chemotherapy regimens as per local institutional protocols either concurrently with or sequentially to trastuzumab.
  Interventions: Biological: trastuzumab; Drug: parenteral chemotherapy
- Arm II (Experimental): Patients receive trastuzumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 6 months in the absence of disease progression or unacceptable toxicity. All patients also receive standard chemotherapy regimens as per local institutional protocols either concurrently with or sequentially to trastuzumab.
  Interventions: Biological: trastuzumab; Drug: parenteral chemotherapy

INTERVENTIONS:
Biological: trastuzumab — Given IV
Drug: parenteral chemotherapy — per the local institutional protocols either concurrently with or sequentially to trastuzumab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known which regimen of trastuzumab is more effective in treating early breast cancer.

PURPOSE: This randomized phase III trial is comparing two trastuzumab regimens to see how well they work in treating women with HER2-positive early breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine disease-free survival of women with HER2-positive early breast cancer treated with neoadjuvant or adjuvant trastuzumab (Herceptin®) for 6 months versus 12 months.

Secondary

* Determine the overall survival of patients treated with these regimens.
* Determine the expected incremental cost effectiveness (cost per quality adjusted life year gained) for 6 months versus 12 months trastuzumab.
* Determine cardiac function as assessed by left ventricular ejection fraction every 3 months during treatment.
* Analyze the predictive factors for development of cardiac damage.

OUTLINE: This is a multicenter study. Patients are stratified according to estrogen receptor status (negative vs positive); chemotherapy timing (adjuvant vs neoadjuvant); chemotherapy type (anthracycline based [no taxane] vs taxane and anthracyclines vs taxane-based [no anthracyclines]); and trastuzumab (Herceptin®) timing (concurrently vs sequentially [with respect to chemotherapy]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive trastuzumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 12 months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive trastuzumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 6 months in the absence of disease progression or unacceptable toxicity.

All patients also receive standard chemotherapy regimens as per local institutional protocols either concurrently with or sequentially to trastuzumab.

Patients complete quality of life questionnaires using the EuroQoL-5D (EQ-5D) at baseline and periodically during study treatment. Patients also complete a diary on out-of-pocket expenses associated with their condition (i.e., travel expenses, over-the-counter medicines and supplements, complementary therapies not funded by NHS, home help, and time away from work) for cost-effective analysis.

After completion of study therapy, patients are followed every 3 months for 1 year, then every 6 months for 1 year, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer
* No evidence of metastatic disease
* Overexpression of HER2 receptor defined as 3+ or 2+ HER2 positivity measured by fluorescent in situ hybridization (FISH) gene amplification
* Indication for chemotherapy based on the following clinical and histopathological features:

  * Receiving or scheduled to receive neoadjuvant chemotherapy

    * Time between diagnosis biopsy and start date of chemotherapy should be less than 1 month
  * Receiving or scheduled to receive adjuvant chemotherapy

    * Completely resected disease, with negative surgical margins (apart from deep margin if full thickness resection)
    * Marginally resected disease and/or positive sentinel nodes allowed provided patients undergo completion of surgery (breast and/or axillary clearance) after chemotherapy
* Hormone receptor status known

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-1
* Adequate bone marrow, hepatic, and renal function
* LVEF normal by ECHO or MUGA
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No clinically significant cardiac abnormalities
* No myocardial infarction within the past 6 months
* No uncontrolled or malignant hypertension
* No history of atrioventricular arrhythmia and/or congestive heart failure (even under medical control), or active second or third degree cardiac block
* No history of allergy to drugs containing polysorbate 20 and the excipient polysorbate 80 (TWEEN 80®) or history of allergy to mouse proteins
* No co-morbidity significantly adding to risks associated with cytotoxic chemotherapy (i.e., severe chronic obstructive pulmonary disease or poorly controlled diabetes)
* No prior diagnosis of malignancy unless managed by surgical treatment only and disease-free for 10 years

  * Prior basal cell carcinoma, cervical carcinoma in situ, or ductal carcinoma in situ of the breast allowed if treated by surgery only
* No concomitant medical or psychiatric problems that might preclude completion of treatment or follow-up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or radiotherapy
* Concurrent radiotherapy allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2007-10; Primary Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival

SECONDARY OUTCOMES:
Overall survival
Cost effectiveness and quality of life
Cardiac function and analysis of predictive factors for development of cardiac damage

CONTACTS AND LOCATIONS:
Overall Officials: Helena Earl, MBBS, PhD, FRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (11):
- United Kingdom (11):
  - Addenbrooke's Hospital, Cambridge, England
  - Cumberland Infirmary, Carlisle, England
  - Derbyshire Royal Infirmary, Derby, England
  - Eastbourne District General Hospital, Eastbourne, England
  - Luton and Dunstable Hospital, Luton, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Peterborough Hospitals Trust, Peterborough, England
  - New Cross Hospital, Wolverhampton, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland

REFERENCES:
- [Derived] Earl H, Hiller L, Vallier AL, Loi S, McAdam K, Hughes-Davies L, Rea D, Howe D, Raynes K, Higgins HB, Wilcox M, Plummer C, Mahler-Araujo B, Provenzano E, Chhabra A, Gasson S, Balmer C, Abraham JE, Caldas C, Hall P, Shinkins B, McCabe C, Hulme C, Miles D, Wardley AM, Cameron DA, Dunn JA. Six versus 12 months' adjuvant trastuzumab in patients with HER2-positive early breast cancer: the PERSEPHONE non-inferiority RCT. Health Technol Assess. 2020 Aug;24(40):1-190. doi: 10.3310/hta24400. PMID 32880572
- [Derived] Earl HM, Hiller L, Vallier AL, Loi S, McAdam K, Hughes-Davies L, Harnett AN, Ah-See ML, Simcock R, Rea D, Raj S, Woodings P, Harries M, Howe D, Raynes K, Higgins HB, Wilcox M, Plummer C, Mansi J, Gounaris I, Mahler-Araujo B, Provenzano E, Chhabra A, Abraham JE, Caldas C, Hall PS, McCabe C, Hulme C, Miles D, Wardley AM, Cameron DA, Dunn JA; PERSEPHONE Steering Committee and Trial Investigators. 6 versus 12 months of adjuvant trastuzumab for HER2-positive early breast cancer (PERSEPHONE): 4-year disease-free survival results of a randomised phase 3 non-inferiority trial. Lancet. 2019 Jun 29;393(10191):2599-2612. doi: 10.1016/S0140-6736(19)30650-6. Epub 2019 Jun 6. PMID 31178152